CLINICAL TRIAL: NCT01947673
Title: Sympathetic Regulation in Intradialytic Hypertension
Brief Title: Mechanisms of Intradialytic Hypertension
Acronym: MID-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Satellite Healthcare (Other)
Responsible Party: Principal Investigator, Jeanie Park, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00066932; 00025948 (Other: Emory)
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Haemodialysis-induced Symptom; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Mindfulness Based Stress Reduction (MBSR) Program (Experimental): After individual instruction, participants in this arm will perform meditation by following a series of mindfulness meditation (MM) recordings during hemodialysis for the next 4 to 8 weeks.The MM instructor will also meet with the participants weekly to provide continued instruction. Participants will also be encouraged to perform MM using a digital audio (MP3) player at home on non-dialysis days, and asked to keep a log of these sessions.
  Interventions: Other: Mindfulness Meditation
- Health Education (Placebo Comparator): Participants randomized to the control condition will undergo a 4 to 8 week health education series, with a parallel protocol as the MBSR intervention. Monitoring of adherence will be same as above.
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Mindfulness Meditation
  Arms: Modified Mindfulness Based Stress Reduction (MBSR) Program
Other: Health Education
  Arms: Health Education

SUMMARY:
Patients with end-stage renal disease (ESRD) are at significantly higher risk for death due to cardiovascular disease. Those with paradoxical increases in blood pressure (BP) during hemodialysis (HD), defined as intradialytic hypertension (IDH), are at even greater risk of cardiovascular mortality. This study seeks to determine the mechanisms that underlie IDH, and whether mindfulness meditation might improve BP during dialysis in these patients. The investigators will first determine if increased adrenaline levels during volume removal contributes to IDH. The investigators will then determine lack of suppression of adrenaline levels in the setting of a high BP also contributes to IDH. This will be done by manipulating blood pressure by using small amounts of vasoactive drugs, and determining if an appropriate response in adrenaline levels occurs. Lastly, the investigators will determine if an intradialytic mindfulness meditation program improves BP and adrenaline levels in ESRD patients with IDH.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients on maintenance hemodialysis for at least 6 months, with increased blood pressure during hemodialysis

Exclusion Criteria:

* drug or alcohol abuse
* any serious systemic disease that might influence survival
* severe anemia with hgb level <8 g/dL
* clinical evidence of congestive heart failure
* ejection fraction below 35%
* myocardial infarction or cerebrovascular accident within the past six months
* symptomatic heart disease determined by electrocardiogram, stress test, and/or history
* treatment with central alpha agonists or monoamine oxidase (MAO) inhibitors
* peripheral neuropathy
* autonomic dysfunction
* pregnancy
* surgery within the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Blood Pressure during dialysis | 8 weeks
Cardiopulmonary baroreflex Sensitivity | 8 weeks

SECONDARY OUTCOMES:
Kidney Disease Quality of Life (KDQOL) Symptom Score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, MD, MS, Principal Investigator — Emory University
Locations (1):
- Emory Dialysis Clinics, Atlanta, Georgia, United States